CLINICAL TRIAL: NCT02702674
Title: The Effect of Coadministration of Oral Propranolol to Oxytocin on Induction of Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: propranolol
Record Dates: First submitted 2016-02-13; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Poor; Labor
MeSH Terms: interventions — Propranolol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propranolol plus oxytocin (Active Comparator): 121 patients who will receive a capsule containing 20 mg propranolol (propranolol plus oxytocin) administrated orally before beginning induction and repeated after 8 hours if no sufficient uterine contractions reached.
  Interventions: Drug: propranolol; Drug: Oxytocin
- placebo plus oxytocin (Placebo Comparator): 121 control patients who will receive a similar capsule as a placebo (oxytocin plus placebo) before beginning induction.
  Interventions: Drug: placebo; Drug: Oxytocin

INTERVENTIONS:
Drug: propranolol — propranolol 20 mg given before induction of labor
  Other Names: indral
  Arms: propranolol plus oxytocin
Drug: placebo — starch tablet containing no active drug material given before induction of labor
  Arms: placebo plus oxytocin
Drug: Oxytocin — intravenous infusion of oxytocin
  Other Names: syntocinon

SUMMARY:
The effect of coadministration of oral propranolol to oxytocin on induction of labor.

DETAILED DESCRIPTION:
Study hypothesis:

Oral propranolol when used with oxytocin during the process of labor may reduce labor interval and decrease the rate of cesarean delivery.

Study population:

The patients will be recruited from the women attending obstetrics reception room, in Ain Shams University Maternity Hospital.

Intervention:

After taking informed consent, all patients recruited in the study will undergo complete clinical examination and detailed medical history will be obtained along with necessary laboratory investigations and ultrasound. Each patient will have a case record form in which the following data will be recorded:

1. History: personal (age, duration of marriage), present illness (any current medical or surgical diseases and any current medication), obstetric history (including parity, gestational age, obstetric complications) and past medical history(especially cardiac problems).
2. Clinical examination:

   1. General examination: assessment of vital data, cardiac and chest auscultation to exclude contraindications for drug administration.
   2. Abdominal examination: assessment of fundal level and contractions if present.
   3. Pelvic examination: assessment of Bishop score, membrane status and fetal presentation.
3. Investigations:

   1. Routine investigations will be done e.g., Full blood count, CRP titre.
   2. Pelvi-abdominal U/S (confirm fetal life, placental location, fetus parameters, amniotic fluid index, expected fetal weight).

Steps:

1. Informed consent will be obtained from parents or guardians of patients who are invited to participate in the research after explanation of benefits and risks of this trial.
2. A capsule containing 20 mg propranolol to the first group (propranolol plus oxytocin) and a similar capsule as a placebo to the second group (oxytocin plus placebo) are administrated orally before beginning induction. Oral capsules are repeated after 8 h, if three forceful contractions are not obtained during 10 min.
3. Induction will be initiated with a dose of 2 mIu/min and increased by 2 mIu/min every 15 min until three forceful contractions be obtained for 10 min, or to a maximum dose of 30 mIu/min. Then, continue at this rate for 8 h. If patients entered the active phase of labor (cervical dilatation = 3-4 cm), induction continue until delivery.
4. Amniotomy is performed when cervical dilation reached 5 cm, if the membrane has not been ruptured spontaneously.
5. The partogram will be used to monitor the fetal heart rate, membrane status, cervical dilation and effacement, station of the fetus, uterine contractions, maternal pulse, maternal blood pressure, maternal temperature.
6. If there is no response to induction on the second day, a cesarean section will be performed.
7. The participants are followed up until delivery.

Safety Considerations:

If the parturient has hyperstimulation of contractions (in a situation with more than 5 contractions/10 min, duration of contraction > 90 sec, interval of contraction less than 2 min, or fetal distress), the induction will be stopped, and the parturient is kept in left lateral position and given oxygen, and intravenous dextrose.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age above 37 weeks.
2. Fetal life positive on ultrasound.
3. Bishop score > 5.
4. Primiparous women.

Exclusion Criteria:

1. history of uterine surgery
2. polyhydramnios
3. contraindications to β-adrenergic agents, such as systolic blood pressure less than 100 mmHg or pulse rate less than 60/min and more than 120/min
4. history of any known cardiac disease
5. mother's pulmonary or metabolic disorders
6. fetal distress
7. estimated weight of the fetus more than 4 kg by ultrasound of cephalic presentation

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 242 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
duration of first stage of labour | 24 hours
  duration of first stage of labour in hours

SECONDARY OUTCOMES:
rate of cesarean section | 48 hours
  number of participants eventually undergo cesarean section
Apgar score | 24 hours
  Apgar score at minute 1 and minute 5 following delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided